CLINICAL TRIAL: NCT04489602
Title: Translation and Validation of the French Version of the ObsQoR-10 Questionnaire for the Evaluation of Recovery After Childbirth: the ObsQoR-10F Questionnaire
Brief Title: Translation and Validation of the French Version of the ObsQoR-10 Questionnaire
Acronym: ObsQoR-10F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: ObsQoR-10F
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Delivery; Childbirth; Patient Reported Outcome Measures; Labor Complication; Quality of Recovery
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Each patient complete ObsQoR-10F questionnaire 3 times (before delivery, on Day 1, on Day 2)
  Interventions: Other: ObsQoR-10F Questionnaire

INTERVENTIONS:
Other: ObsQoR-10F Questionnaire — The ObsQoR-10F questionnaire consists of 10 items assessing different aspects of postpartum recovery: physical comfort and pain, physical independence and emotional status. It takes two minutes to complete all the items. If the patient is not able to read the questionnaire herself, a third person can ask the questions orally to the patient. If the patient has returned home with her child, she can be contacted by phone to complete the questionnaire. Each item is scored from 0 to 10 and the total score is the sum of the score for each item, which is a score from 0 to 110.

SUMMARY:
Until recently, there was no validated scoring tool to assess recovery after childbirth. Ciechanowicz et al. developed and validated a postpartum recovery score for women with a caesarean section (scheduled or unscheduled): the ObsQoR-11. The psychometric validation of the ObsQoR-11 confirms its reliability, its response to change, its acceptability and its feasibility (average filling time of 2 minutes, and the possibility to print the questionnaire on one page). The use of this score allows the investigators to quantify the quality of the patient's recovery between 0 and 110 (0 being a really poor recovery, and 110 a total recovery), by allocating a score from 0 to 10 for each item.

Since then, the initial version of ObsQoR-11 has evolved into a smaller version, ObsQoR-10, for which the pain items have been merged. Similarly, by assigning a score from 0 to 10 for each item, the ObsQoR-10 score allows to quantify the quality of the patient's recovery between 0 and 100 (0 being a very poor recovery, and 100 being full recovery).

There are currently no translations of this score into another language, but the investigators can easily assume that they will be done in the near future. French remains the fifth most spoken language in the world. The investigators therefore feel it is necessary to validate the translated version of the ObsQoR-10 score.

DETAILED DESCRIPTION:
Recovery after childbirth (by caesarean section or vaginal delivery) is a complex process, depending on the characteristics of the patient, the anaesthesia, and the need for surgery or an instrumental device. This event is a source of stress, anxiety and pain, and can also lead to postpartum complications. Studies evaluating interventions during childbirth traditionally focus on mortality and morbidity which, although important, do not describe the patient's experience or the quality of her recovery.

Scores for measuring the quality of post-operative recovery have been developed. These scoring tools accurately measure post-operative recovery by looking at some dimensions of the patient's experience. However, they have been developed and validated in non-obstetrical patients. They therefore contain aspects of recovery that are not relevant to delivery and postpartum. Furthermore, they do not include key elements, such as the ability to care for the newborn.

Until recently, there was no validated scoring tool to assess recovery after childbirth. Ciechanowicz et al. developed and validated a postpartum recovery score for women with a caesarean section (scheduled or unscheduled): the ObsQoR-11. This multidimensional score is a questionnaire of 11 items evaluating: moderate pain, severe pain, nausea and vomiting, feeling of discomfort, shivering, feeling of comfort, ability to mobilize, ability to carry the newborn, ability to feed, ability to groom alone, and finally feeling of self-control. The psychometric validation of the ObsQoR-11 confirms its reliability, its response to change, its acceptability and its feasibility (average filling time of 2 minutes, and the possibility to print the questionnaire on one page). The use of this score allows to quantify the quality of the patient's recovery between 0 and 110 (0 being a really poor recovery, and 110 a total recovery), by allocating a score from 0 to 10 for each item.

This tool has the advantage of efficiently evaluating the concept of immediate postpartum recovery, with an acceptable feasibility for both the patient and the caregivers. Since then, the initial version of ObsQoR-11 has evolved into a smaller version, ObsQoR-10, for which the pain items have been merged. Similarly, by assigning a score from 0 to 10 for each item, the ObsQoR-10 score allows to quantify the quality of the patient's recovery between 0 and 100 (0 being a very poor recovery, and 100 being full recovery).

There are currently no translations of this score into another language, but the investigators can easily assume that they will be done in the near future. French remains the fifth most spoken language in the world. The investigators therefore feel it is necessary to validate the translated version of the ObsQoR-10 score.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old);
* French-speaking;
* Admitted for spontaneous obstetrical labor, induction of obstetrical labor, or scheduled cesarean section;
* Able to answer the questionnaire, alone or with the help of a third party;
* Agreeing to participate in the study

Exclusion Criteria:

* Psychiatric or neurological pathology compromising cooperation in the questionnaire validation protocol,
* Psychological history (medical termination of pregnancy, foetal death in utero).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for spontaneous obstetrical labor, induction of obstetrical labor, or scheduled cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Validity of ObsQoR-10F questionnaire | 2 days
  Evaluate the validity of the French version of the ObsQoR-10 to assess immediate postpartum recovery (at 24 and 48 hours after vaginal delivery or Caesarean section).

SECONDARY OUTCOMES:
Validity of ObsQoR-10F questionnaire (Caesarean section) | 2 days
  Ensure the validity of the questionnaire in the sub-population of Caesarean delivery population (scheduled and unscheduled) at 24 and 48 hours

OTHER OUTCOMES:
Validity of ObsQoR-10F questionnaire (Vaginal delivery) | 2 days
  Assess the validity of the questionnaire specifically in the subpopulation of patients with a vaginal delivery (with or without instrumental extraction) at 24 and 48 hours
Minimal important difference | 2 days
  Estimate minimal important difference from the ObsQoR-10F questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Background] Sultan P, Kormendy F, Nishimura S, Carvalho B, Guo N, Papageorgiou C. Comparison of spontaneous versus operative vaginal delivery using Obstetric Quality of Recovery-10 (ObsQoR-10): An observational cohort study. J Clin Anesth. 2020 Aug;63:109781. doi: 10.1016/j.jclinane.2020.109781. Epub 2020 Mar 20. PMID 32203873
- [Derived] Mazoue E, Veret M, Corroenne R, Mercier MB, Lomo H, Verhaeghe C, Lasocki S, Bouet PE, Leger M. Translation and validation of the French version of the ObsQoR-10 questionnaire for the evaluation of recovery after delivery: the ObsQoR-10-French. BJA Open. 2023 Aug 17;7:100221. doi: 10.1016/j.bjao.2023.100221. eCollection 2023 Sep. PMID 37638079